CLINICAL TRIAL: NCT03494400
Title: Effects of Aerobic Training in Treatment for Breast Cancer
Brief Title: Aerobic Training in Treatment for Breast Cancer
Acronym: ATTBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Andréa Dias Reis, Clinical Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: State University of São Paulo
Record Dates: First submitted 2018-03-14; First posted 2018-04-11 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Cancer of Breast; Healthy
Keywords: Breast cancer; Physical exercise; Body mass
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Presential Aerobic Training with Hormone Therapy (Experimental): A group of women with breast cancer who use Tamoxifen or Aromatase Inhibitor and will perform presential aerobic training.
  Interventions: Other: Aerobic Training Presential
- Presential Aerobic Training without Breast Cancer (Active Comparator): A group of women without breast cancer who use Aromatase Inhibitor and will perform presential aerobic training.
  Interventions: Other: Aerobic Training Presential
- Home-based Aerobic Training with Hormone Therapy (Experimental): A group of women with breast cancer who use Tamoxifen or Aromatase Inhibitor and will perform home-based aerobic training.
  Interventions: Other: Aerobic Training Home-based
- Home-based Aerobic Training without Breast Cancer (Active Comparator): A group of women without breast cancer who use Aromatase Inhibitor and will perform aerobic training home-based.
  Interventions: Other: Aerobic Training Home-based

INTERVENTIONS:
Other: Aerobic Training Presential — The intervention will last 24 weeks, in which the presential training group will undergo aerobic training three times a week on interspersed days, more follow-up.
  Other Names: Physical exercise Presential
  Arms: Presential Aerobic Training with Hormone Therapy; Presential Aerobic Training without Breast Cancer
Other: Aerobic Training Home-based — The intervention will last 24 weeks, the group accompanied by the distance will carry out the activities in their preferred place under the distance supervision of professionals and every 14 days must attend the UNESP to adjust the intensity and verification of attendance to the proposed activities, more follow-up.
  Other Names: Physical exercise Home-based
  Arms: Home-based Aerobic Training with Hormone Therapy; Home-based Aerobic Training without Breast Cancer

SUMMARY:
Introduction. Treatment with hormone therapy reduced the likelihood of tumor recurrence and metastasis in the patient. However, it has adverse effects such as: loss of bone mineral density, increase in body weight, metabolic changes and, consequently, lower quality of life. Physical training has been used as a means of reducing these and other adverse effects, but there is no definite protocol on which training model is effective, especially in patients who only use Tamoxifen or Aromatase Inhibitor as an adjuvant therapy for treatment of breast cancer.

Objective: To compare the effect of aerobic training on body composition, metabolic and inflammatory variables, physical activity level, sleep, anxiety, depression, body image, fatigue, strength, flexibility and quality of life of women undergoing breast cancer treatment use Tamoxifen and Aromatase Inhibitor and women without cancer.

Method. The sample will be formed by women without cancer and under treatment with hormone therapy being accompanied by the public service for treatment of breast cancer of the city of Presidente Prudente. A 24-week notification in which the face-to-face training group will undergo aerobic training three times a week on interspersed days and the group accompanied at a distance will perform as a preferred activity under a distance supervision of professionals every 14 days of return to attend the UNESP for the adequacy of the analysis and selection of attendance to the proposed activities. Evaluations of the variables of interest at the baseline of the intervention will be performed after 12 weeks and soon after the intervention. The investigators will analyze: biomarkers (TNFα, LDL, HDL, VLDL, as well as in the lipid profile (triglycerides, total cholesterol and LDL fractions ), glycemia, insulin, anthropometric measurements, physical activity level, sleep, pain, anxiety, depression, body image, fatigue, strength, flexibility. Trainings will be performed within the target zone of maximum heart rate. Comparisons between groups at each time point will be performed using Student's T-test for independent samples. The comparisons of the variables of interest at the initial moment and after 12 and 24 weeks will be made through the multivariate analysis, where the group effects, time and interaction of both will be compared. All analyzes will be performed in SPSS software version 24.0 and significance of 5%.

DETAILED DESCRIPTION:
Introduction. Breast cancer is one of the leading causes of morbidity and mortality in the world.Treatment with hormone therapy reduced the likelihood of tumor recurrence and metastasis in the patient. However, it has adverse effects such as: loss of bone mineral density, increase in body weight, metabolic changes (lipid and low grade systemic inflammation) and, consequently, lower quality of life. Physical training has been used as a means of reducing these and other adverse effects, but there is no definite protocol on which training model is effective, especially in patients who only use Tamoxifen or Aromatase Inhibitor as an adjuvant therapy for treatment of breast cancer.

Objective: To compare the effect of aerobic training on body composition, metabolic and inflammatory variables, physical activity level, sleep, anxiety, depression, body image, fatigue, strength, flexibility and quality of life of women undergoing breast cancer treatment use Tamoxifen and Aromatase Inhibitor and women without cancer.

Method. The sample will be formed by women without cancer and under treatment with hormone therapy being accompanied by the public service for treatment of breast cancer of the city of Presidente Prudente. Where participants will be distributed in six groups submitted to intervention with aerobic training: Tamoxifen group with face-to-face training (GTP); Aromatase Inhibitor Group with face-to-face training (GIP); Tamoxifen training group by distance monitoring (GTA); Training group Aromatase inhibitor by distance monitoring (GIA); Group without training with cancer (GC) and Group training face-to-face without cancer (GTSC). A 24-week notification in which the face-to-face training group will undergo aerobic training three times a week on interspersed days and the group accompanied at a distance will perform as a preferred activity under a distance supervision of professionals every 14 days of return to attend the UNESP for the adequacy of the analysis and selection of attendance to the proposed activities. Evaluations of the variables of interest at the baseline of the intervention will be performed after 12 weeks and soon after the intervention. The investigators will analyze: biomarkers will analyze: biomarkers (Tumor Necrosis Factor-Alpha (TNFα), (LDL), High Density Lipoprotein (HDL), and Very Low Density Lipoprotein (VLDL), as well as in the lipid profile (triglycerides, total cholesterol and low density lipoprotein (LDL) fractions) ), glycemia, insulin, anthropometric measurements, physical activity level, sleep, pain, anxiety, depression, body image, fatigue, strength, flexibility. Trainings will be performed within the target zone of maximum heart rate. Comparisons between groups at each time point will be performed using Student's T-test for independent samples. The comparisons of the variables of interest at the initial moment and after 12 and 24 weeks will be made through the multivariate analysis, where the group effects, time and interaction of both will be compared. All analyzes will be performed in SPSS software version 24.0 and significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer;
* Perform Tamoxifen or Aromatase Inhibitor Treatment;
* Being in stages 1 to 3 of breast cancer;
* Do not present physical limitations or any health problem that prevents the performance of the evaluations and the training;
* Have a medical certificate to perform the ergometric test and participate in physical training;
* Not practicing physical training in the last six months;
* Sign the Term of Free Consent and Clarification.

Inclusion Criteria for the group without cancer

* Do not use Tamoxifen or Aromatase Inhibitor;
* Not being diagnosed with any type of cancer.

Exclusion Criteria:

* Accumulate three consecutive absences or four non-consecutive absences in presential training during the month;
* Failure to attend the scheduled bi-weekly activities in the case of the home-based training group;
* Do not send information about the activities carried out in the case of the home-based group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of body composition by Bone Densitometry (DEXA) equipment | 24 week
  Reduction of body mass and of increased fat free mass

SECONDARY OUTCOMES:
Evaluation of quality of life by questionnarie EORTC-QLQ-30 | 24 week
  Increased of quality of life global
Evaluation inflammatory response by ELISA equipment | 24 week
  Reduction of interleukin- IL 6
Evaluation of pain by questionnarie BPI. | 24 week
  Reduction of pain intensity to increased of functional capacity
Evaluation of level of physical activity by triaxial accelerometer equipment | 24 week
  Increased of level of physical activity
Nutritional evaluation by food register | 24 week
  Increased of quality of food

CONTACTS AND LOCATIONS:
Overall Officials: ISMAEL F FREITAS JUNIOR, Study Director — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- Faculdade de Ciências e Tecnologia, Universidade Estadual Paulista Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battaglini CL, Mills RC, Phillips BL, Lee JT, Story CE, Nascimento MG, Hackney AC. Twenty-five years of research on the effects of exercise training in breast cancer survivors: A systematic review of the literature. World J Clin Oncol. 2014 May 10;5(2):177-90. doi: 10.5306/wjco.v5.i2.177. PMID 24829866
- [Background] Do J, Cho Y, Jeon J. Effects of a 4-week multimodal rehabilitation program on quality of life, cardiopulmonary function, and fatigue in breast cancer patients. J Breast Cancer. 2015 Mar;18(1):87-96. doi: 10.4048/jbc.2015.18.1.87. Epub 2015 Mar 27. PMID 25834616
- [Background] Eriksen AK, Hansen RD, Borre M, Larsen RG, Jensen JM, Overgaard K, Borre M, Kyro C, Landberg R, Olsen A, Tjonneland A. A lifestyle intervention among elderly men on active surveillance for non-aggressive prostate cancer: a randomised feasibility study with whole-grain rye and exercise. Trials. 2017 Jan 13;18(1):20. doi: 10.1186/s13063-016-1734-1. PMID 28086943
- [Background] Nyrop KA, Callahan LF, Rini C, Altpeter M, Hackney B, Schecher A, Wilson A, Muss HB. Adaptation of an Evidence-Based Arthritis Program for Breast Cancer Survivors on Aromatase Inhibitor Therapy Who Experience Joint Pain. Prev Chronic Dis. 2015 Jun 11;12:E91. doi: 10.5888/pcd12.140535. PMID 26068412
- [Background] Travier N, Velthuis MJ, Steins Bisschop CN, van den Buijs B, Monninkhof EM, Backx F, Los M, Erdkamp F, Bloemendal HJ, Rodenhuis C, de Roos MA, Verhaar M, ten Bokkel Huinink D, van der Wall E, Peeters PH, May AM. Effects of an 18-week exercise programme started early during breast cancer treatment: a randomised controlled trial. BMC Med. 2015 Jun 8;13:121. doi: 10.1186/s12916-015-0362-z. PMID 26050790